CLINICAL TRIAL: NCT00520130
Title: Phase II Trial of Targeted Immune-Depleting Chemotherapy and Reduced-Intensity Allogeneic Hematopoietic Stem Cell Transplantation Using 8/8 and 7/8 HLA-matched Unrelated Donors and Utilizing Two Graft-versus-Host Disease Prophylaxis Regimens for the Treatment of Leukemias, Lymphomas, and Pre-malignant Blood Disorders
Brief Title: Chemotherapy and Unrelated Donor Stem Cell Transplantation for Patients With Cancers of the Blood and Immune System
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Pavletic, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070195; 07-C-0195
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Myelodysplastic Syndrome; Hodgkin's Lymphoma; Non-Hodgkin's Disease; Acute Leukemia; Multiple Myeloma
Keywords: Unrelated Donors; Reduced Intensity Stem Cell Transplant; Leukemia; Lymphoma; Allogeneic Stem Cell Transplant; Myelodysplastic Syndrome; Multiple Myeloma
MeSH Terms: conditions — Myelodysplastic Syndromes; Hodgkin Disease; Multiple Myeloma; Leukemia; Lymphoma | interventions — Rituximab; Cyclosporine; Tacrolimus; Filgrastim; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A - Tacrolimus, methotrexate, sirolimus (TMS) Arm (Experimental): TMS Arm
  Interventions: Biological: Rituximab; Drug: Allogenic stem cell transplant (ASCT); Drug: Conditioning Chemotherapy; Drug: TMS; Drug: FLAG; Drug: EPOCH-F
- B - Cyclosporine (AC) Arm (Experimental): AC Arm
  Interventions: Biological: Rituximab; Drug: Cyclosporine; Drug: Allogenic stem cell transplant (ASCT); Drug: Conditioning Chemotherapy; Drug: FLAG; Drug: EPOCH-F; Biological: Alemtuzumab

INTERVENTIONS:
Biological: Rituximab — Rituximab: 375 mg/m(2) intravenous (IV), day 1 for patients with cluster of differentiation 20 (CD20)-positive disease.
  Other Names: Rituxan
Drug: Cyclosporine — Cyclosporine: IV over 2 hours or orally every 12 hours on days -1 to 100, followed by a taper if graft versus host disease (GVHD) does not develop.
  Other Names: Neoral
  Arms: B - Cyclosporine (AC) Arm
Drug: Allogenic stem cell transplant (ASCT) — Allogenic stem cell transplant
Drug: Conditioning Chemotherapy — Fludarabine:30 mg/m(2) per day IV infusion over 30 minutes, daily. On days -6, -5, -4, and -3.
  Cyclophosphamide:1200 mg/m(2) per day IV infusion over 2 hours on Days 6, -5, -4, -3 Mesna: 1200 mg/m(2) per day IV infusion, Daily on days 6, -5,-4, and -3
Drug: TMS — Tacrolimus: starting day -3 before transplant, given initially at 0.02 mg/kg/day CIV. Continue IV and then switch to an equivalent oral dose (when patient taking po) titrated for a goal level of 5 to 10 ng/ml; Sirolimus: given as an initial loading dose of 12 mg p.o. on day -3 pre-transplant, 4 mg starting day -2 pre-transplant and titrated for levels 3-12 ng/ml; Methotrexate 5 mg/m2 IV on days +1, +3, +6, and +11 post-transplant. Tacrolimus and sirolimus will be tapered at day +63, day +119 and day +180 post-transplant as tolerated.
  Other Names: Prograf
  Arms: A - Tacrolimus, methotrexate, sirolimus (TMS) Arm
Drug: FLAG — Fludarabine:25 mg/m(2) per day IV over 30 minutes, Daily on days 1-5 Cytarabine: 2,000 mg/m(2) IV over 4 hours,on Days 1, 2, 3, 4, 5 Filgrastim: 5 mcg/kg per day subcutaneous (SC) beginning 24 hours PRIOR to initiation of chemotherapy
  Other Names: Fludarabine+high-dose cytarabine+G-CSF (Filgrastim))
Drug: EPOCH-F — Fludarabine:25 mg/m(2) per day IV infusion over 30 minutes, daily on days 1-4 Etoposide :50 mg/m(2) per day continuous IV infusion over 24 hours on days 1-4 Doxorubicin:10 mg/m(2)/day CIV, days 1-4 Vincristine:0.4 mg/m(2) per day continuous IV infusion over 24 hours daily on days 1-4 Cyclophosphamide:750 mg/m(2) IV infusion over 30 minutes on day 5
Biological: Alemtuzumab — Alemtuzumab:20 mg/day IV over 8 h on days 8 to 4 pre-transplant.
  Other Names: Campath
  Arms: B - Cyclosporine (AC) Arm

SUMMARY:
Background:

Major problems with stem cell transplantation (SCT) for cancer treatment are a lack of suitable donors for patients without a human leukocyte-antigen (HLA) tissue-matched sibling and graft-versus-host disease (GVHD), a serious side effects of immune-suppressing chemotherapy that is given to bring the cancer under control before SCT. In GVHD, the patients immune system attacks the transplanted donor cells.

This study will try to improve the results of SCT from unrelated HLA-matched donors using targeted immune-depleting chemotherapy to bring the cancer under control before transplantation and to lower the chance of graft rejection, followed by reduced-intensity transplant chemotherapy to make the procedure less toxic.

Objectives:

To evaluate the safety and effectiveness of targeted immune-depleting chemotherapy followed by reduced-intensity transplant chemotherapy in patients with advanced cancers of the blood and immune system.

To evaluate the safety and effectiveness of two different drug combinations to prevent GVHD. Both regimens have been successful in preventing GVHD, but they work by different mechanisms and affect the rebuilding of the immune system after the transplant.

Eligibility:

People 18 to 74 years of age with advanced or high-risk cancers of the blood and immune system who do not have a suitable HLA-matched sibling.

Design:

All patients receive chemotherapy before transplant to treat the cancer and suppress immune function.

All patients receive a conditioning regimen of cyclophosphamide for 4 days and fludarabine for 4 days before SCT to prepare for the transplant.

Patients are randomly assigned to one of two combination drug treatments to prevent GHVD as follows:

* Group 1: Tacrolimus starting 3 days before SCT and continuing for 6 months, plus methotrexate on days 1, 3, 6, and 11 post-SCT, plus sirolimus starting 3 days before the SCT and continues for 6 months following SCT.
* Group 2: Alemtuzumab for 4 days starting 8 days before SCT, plus cyclosporine starting 1 day before SCT and continuing for 6 months.

Patients receive the donors stem cells and immune cells 2 days after completing the conditioning regimen.

Patients are followed at the clinic regularly for the first 6 months after SCT, and then less often for at least 5 years. Some visits may include bone marrow aspirates and biopsies, blood draws, and other tests to monitor disease status.

A skin biopsy, oral mucosa biopsy, and saliva collection are done to study chronic GVHD.

...

DETAILED DESCRIPTION:
Background:

* The major limitations to the broader applicability of allogeneic hematopoietic stem cell transplantation (HSCT) for the treatment of malignancies are lack of suitable donors and therapy-related toxicities which include delayed and incomplete immune reconstitution and graft-versus-host disease (GVHD). Based on the theory that the rapid establishment of donor chimerism was essential for an optimal graft-versus-tumor effect, we have employed a strategy of targeted immune depleting chemotherapy prior to reduced-intensity allogeneic HSCT. It is our intent to investigate this approach in the setting of human leukocyte-antigen (HLA)-matched unrelated donors in a pilot manner.
* A clearly superior GVHD prophylaxis regimen has not been established in the unrelated donor transplant setting. The best results that have been reported are with the combination of alemtuzumab plus cyclosporine [AC] and the combination of tacrolimus, methotrexate, and sirolimus [TMS]. These two regimens work by mechanisms which are biologically distinct and potentially have markedly different effects upon immune reconstitution that have not been well studied. In addition, neither of these regimens has been assessed for their effects on chronic GVHD using the National Institutes of Health (NIH) Consensus Conference Criteria. It is our intent to study the effects that these two regimens have on immune reconstitution and chronic GVHD in the setting sequential targeted immune-depleting chemotherapy and reduced-intensity allogeneic HSCT from HLA-matched unrelated donors.

Objectives:

* Primary objectives:

  1. to assess the effects of two biologically distinct GVHD prophylaxis regimens, TMS and AC, on immune reconstitution in patients receiving targeted-immune depletion and reduced-intensity allogeneic HSCT from HLA-matched unrelated donors. As part of a comprehensive assessment of immune reconstitution, the primary immunologic endpoint will be the determination of cluster of differentiation 4 (CD4)+ T cell receptor V BETA repertoire by complementarity determining region 3 (CDR3) spectratyping at 3 months post-transplant.
  2. to assess overall safety of these two regimens in this setting, as determined by engraftment, acute GVHD, early and late treatment-related mortality, and overall survival.
  3. to determine and monitor incidence, organ severity and overall severity of chronic GVHD prospectively using the newly developed NIH Consensus Conference diagnosis and staging criteria and preliminarily validate those tools for use in clinical practice and trials.
* Secondary objectives include further assessment of immune reconstitution, study of engraftment kinetics, and assessment of those patients who receive higher doses of anthracyclines for long and short term toxicities

Eligibility:

* Adults (18-74 years) with advanced or high risk hematologic malignancies including acute myeloid leukemia (AML), acute lymphocytic leukemia (ALL), myelodysplastic syndrome (MDS), chronic lymphocytic leukemia (CLL), non-hodgkin lymphoma (NHL), hodgkin lymphoma (HL), chronic myelogenous leukemia (CML), multiple myeloma, and myeloproliferative disorder (MPD) who lack a suitable HLA matched sibling.
* An unrelated donor matched at a minimum of 7 of 8 alleles (HLA-A,-B,-C, and DRB1) by high resolution typing, identified through the National Marrow Donor Program.
* Life expectancy of at least 3 months, Eastern Cooperative Oncology Group (ECOG) less than or equal to 2 and relatively normal major organ functions.

Design:

* Patients will receive disease-specific induction chemotherapy (etoposide, prednisone, vincristine, cyclophosphamide and doxorubicin (EPOCH-fludarabine (F)/rituximab (R) or fludarabine, cytarabine, and granulocyte colony-stimulating factor (FLAG)) prior to transplant for disease control and immune depletion. If disease is controlled (greater than partial response (PR)) and immune depletion objectives have been met, patients may forgo induction chemotherapy and move forward to the transplant conditioning regimen.
* All patients will receive an identical conditioning regimen consisting of cyclophosphamide 1200 mg/m(2)/day intravenous (IV) for 4 days and fludarabine 30 mg/m(2)/day for 4 days.
* Patients will be stratified according to degree of HLA-match and randomized at the time of enrollment to one of two GHVD prophylaxis regimens:

  * Group 1: Tacrolimus starting 3 days before stem cell transplant (SCT), and continuing for 6 months, plus methotrexate on days 1, 3, 6, and 11 post-SCT, plus sirolimus starting 3 days before the SCT and continues for 6 months following SCT.
  * Group 2: Alemtuzumab for 4 days starting 8 days before SCT, plus cyclosporine starting 1 day before SCT and continuing for 6 months.
* A maximum of 105 patients will be enrolled and randomly assigned to the two arms in order to yield 44 patients per arm (88 total patients) who are able to be evaluated for development of severe chronic GVHD.

ELIGIBILITY:
* ELIGIBILITY CRITERIA RECIPIENT ON STANDARD CARE THERAPY:
* The patient is 18-74 years of age.
* The patient has a potentially suitable 8/8 donor if they are between the ages of 69-74 years of age or a potentially suitable 8/8 or 7/8 unrelated donor(s) in the National Marrow Registry or Other Available Registry if they are between the ages of 18-74.
* The patient currently does not meet the protocol s eligibility/enrollment criteria for any reason.
* There is a high likelihood that the patient, in the opinion of the principal investigator (PI) or lead associate investigator (LAI), will meet the protocols eligibility/enrollment criteria to proceed to transplant after standard therapy is completed.
* The patient or legal guardian is able to give informed consent.

EXCLUSION CRITERIA RECIPIENT ON STANDARD CARE THERAPY:

* Human immunodeficiency virus (HIV) infection. There is theoretical concern that the degree of immune suppression associated with the treatment may result in progression of HIV infection.
* Pregnant or lactating. Patients of childbearing potential must use an effective method of contraception. The effects of the chemotherapy, the subsequent transplant and the medications used after the transplant are highly likely to be harmful to a fetus. The effects upon breast milk are also unknown and may be harmful to the infant.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-10-30 (Actual); Primary Completion 2015-10-14 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Z Pavletic, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pavletic SZ, Martin P, Lee SJ, Mitchell S, Jacobsohn D, Cowen EW, Turner ML, Akpek G, Gilman A, McDonald G, Schubert M, Berger A, Bross P, Chien JW, Couriel D, Dunn JP, Fall-Dickson J, Farrell A, Flowers ME, Greinix H, Hirschfeld S, Gerber L, Kim S, Knobler R, Lachenbruch PA, Miller FW, Mittleman B, Papadopoulos E, Parsons SK, Przepiorka D, Robinson M, Ward M, Reeve B, Rider LG, Shulman H, Schultz KR, Weisdorf D, Vogelsang GB; Response Criteria Working Group. Measuring therapeutic response in chronic graft-versus-host disease: National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. Response Criteria Working Group report. Biol Blood Marrow Transplant. 2006 Mar;12(3):252-66. doi: 10.1016/j.bbmt.2006.01.008. PMID 16503494
- [Background] Shaffer BC, Modric M, Stetler-Stevenson M, Arthur DC, Steinberg SM, Liewehr DJ, Fowler DH, Gale RP, Bishop MR, Pavletic SZ. Rapid complete donor lymphoid chimerism and graft-versus-leukemia effect are important in early control of chronic lymphocytic leukemia. Exp Hematol. 2013 Sep;41(9):772-8. doi: 10.1016/j.exphem.2013.04.015. Epub 2013 May 18. PMID 23689118
- [Background] Pavletic SZ, Lee SJ, Socie G, Vogelsang G. Chronic graft-versus-host disease: implications of the National Institutes of Health consensus development project on criteria for clinical trials. Bone Marrow Transplant. 2006 Nov;38(10):645-51. doi: 10.1038/sj.bmt.1705490. Epub 2006 Sep 18. PMID 16980994
- [Background] Hardy NM, Fellowes V, Rose JJ, Odom J, Pittaluga S, Steinberg SM, Blacklock-Schuver B, Avila DN, Memon S, Kurlander RJ, Khuu HM, Stetler-Stevenson M, Mena E, Dwyer AJ, Levine BL, June CH, Reshef R, Vonderheide RH, Gress RE, Fowler DH, Hakim FT, Bishop MR. Costimulated tumor-infiltrating lymphocytes are a feasible and safe alternative donor cell therapy for relapse after allogeneic stem cell transplantation. Blood. 2012 Mar 22;119(12):2956-9. doi: 10.1182/blood-2011-09-378398. Epub 2012 Jan 30. PMID 22289893
- [Derived] Holtzman NG, Curtis LM, Salit RB, Shaffer BC, Pirsl F, Ostojic A, Steinberg SM, Schulz E, Wilder JS, Hughes TE, Rose J, Memon S, Korngold R, Gea-Banacloche JC, Fowler DH, Hakim FT, Gress RE, Bishop MR, Pavletic SZ. High-dose alemtuzumab and cyclosporine vs tacrolimus, methotrexate, and sirolimus for chronic graft-versus-host disease prevention. Blood Adv. 2024 Aug 27;8(16):4294-4310. doi: 10.1182/bloodadvances.2023010973. PMID 38669315
- [Derived] Assmann JC, Farthing DE, Saito K, Maglakelidze N, Oliver B, Warrick KA, Sourbier C, Ricketts CJ, Meyer TJ, Pavletic SZ, Linehan WM, Krishna MC, Gress RE, Buxbaum NP. Glycolytic metabolism of pathogenic T cells enables early detection of GVHD by 13C-MRI. Blood. 2021 Jan 7;137(1):126-137. doi: 10.1182/blood.2020005770. PMID 32785680
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-C-0195.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 89 participants in the study. 3 patients enrolled and their cancers progressed prior to randomization so they were taken off study. 3 of these participants went back into remission with additional chemo and were re-enrolled on the protocol and randomized. They are counted twice in the enrolment (e.g. 92) but only once in the Started row.
Groups:
- A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm: Rituximab: 375 mg/m2 intravenous (IV), day 1 for patients (pts) with cluster of differentiation 20-positive disease. Allogenic stem cell transplant (txplt). Fludarabine:30 mg/m2 per day IV over 30 min. daily. On days -6, -5, -4, and -3. Cyclophosphamide:1200 mg/m2 per day IV over 2 hrs on Days 6, -5, -4, -3. Mesna:1200 mg/m2 per day IV, Daily on days 6, -5,-4, and -3.Tacrolimus: day -3 before txplt, 0.02 mg/kg/day CIV, then switch to an equivalent oral dose (when pts taking po) titrated for a goal level of 5-10 ng/ml; Sirolimus: loading dose of 12 mg p.o. on day -3 pre-txplt, 4 mg day -2 pre-txplt and titrated for levels 3-12 ng/ml; Methotrexate 5 mg/m2 IV on days +1, +3, +6, and +11 post txplt). Tacrolimus and sirolimus will be tapered at day +63, day +119 and day +180 post-txplt as tolerated. Fludarabine:25 mg/m2 per day IV over 30 minutes, Daily on days 1-5.Cytarabine: 2,000 mg/m2 IV over 4 hrs, on Days 1, 2, 3, 4, 5. Filgrastim: 5 mcg/kg per day SC beginning 24 hrs before chemo.
- B - Cyclosporine (AC) Arm: Rituximab375 mg/m2 IV, day 1 for pts with CD20-positive disease. Cyclosporine IV over 2 hrs or orally every 12 hrs on days -1-100, followed by a taper if GVHD does not develop. Allogenic stem cell transplant. Conditioning Chemotherapy Fludarabine:30 mg/m2 per day IV infusion over 30 min., daily on days -6, -5, -4, and -3. Cyclophosphamide1200 mg/m2 per day IV infusion over 2 hrs on Days 6, -5, -4, -3. Mesna1200 mg/m2 per day IV infusion, Daily on days 6, -5,-4, and -3. FLAG: Fludarabine25 mg/m2 per day IV over 30 min., Daily on days 1-5. Cytarabine 2,000 mg/m2 IV over 4 hrs, on Days 1, 2, 3, 4, 5. Filgrastim 5 mcg/kg per day SC beginning 24 hrs PRIOR to start of chemotherapy. EPOCH-F: Fludarabine25 mg/m2 per day IV infusion over 30 min., daily on days 1-4. Etoposide 50 mg/m2 per day continuous IV infusion over 24 hrs on days 1-4. Doxorubicin10 mg/m2/d. Grp 2 Alemtuzumab for 4 days starting 8 days before SCT + cyclosporine starting 1 day before SCT and continuing for 6 months.
Period: Overall Study
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
Started | 44 | 45
Completed | 39 | 44
Not Completed | 5 | 1
Not completed — Disease progression on study | 4 | 0
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: There were 89 participants in the study. 3 patients enrolled and their cancers progressed prior to randomization so they were taken off study. 3 of these participants went back into remission with additional chemo and were re-enrolled on the protocol and randomized. They are counted twice in the enrolment (e.g. 92) but only once in the Started row.
Groups:
- Tacrolimus, Methotrexate, Sirolimus (TMS) Arm: Rituximab:375 mg/m2 IV, day 1 for patients with CD20-positive disease. Allogenic stem cell transplant (ASCT):Conditioning Chemotherapy:Fludarabine:30 mg/m2 per day IV infusion over 30 minutes, daily On days -6, -5, -4, and -3. Cyclophosphamide:1200 mg/m2 per day IV infusion over 2 hours on Days 6, -5, -4, -3.Mesna: 1200 mg/m2 per day IV infusion, Daily on days 6, -5,-4, and -3.Tacrolimus: 0.02 mg/kg, start day 3. Continue IV or PO. Taper will begin at day +63 if no acute GVHD then at day +119 and discontinue at day +180 as tolerated. Methotrexate: 5mg/m2 IV over 15 minutes on days 1, 3, 6, and 11. Sirolimus: 12 mg PO on days -3 to 63, followed by a taper if GVHD does not develop. Sirolimus: 12 mg PO on days -3 to 63, followed by a taper if GVHD does not develop.FLAG: Fludarabine:25 mg/m2 per day IV over 30 minutes, Daily on days 1-5. Cytarabine: 2,000 mg/m2 IV over 4 hours, on Days 1, 2, 3, 4, 5. Filgrastim: 5 mcg/kg per day SC beginning 24 hours PRIOR to initiation of chemotherapy
- Cyclosporine (AC) Arm: Rituximab375 mg/m2 IV, day 1 for pts with CD20-positive disease. Cyclosporine IV over 2 hrs or orally every 12 hrs on days -1-100, followed by a taper if GVHD does not develop. Allogenic stem cell transplant. Conditioning Chemotherapy Fludarabine:30 mg/m2 per day IV infusion over 30 min., daily on days -6, -5, -4, and -3. Cyclophosphamide1200 mg/m2 per day IV infusion over 2 hrs on Days 6, -5, -4, -3. Mesna1200 mg/m2 per day IV infusion, Daily on days 6, -5,-4, and -3. FLAG: Fludarabine25 mg/m2 per day IV over 30 min., Daily on days 1-5. Cytarabine 2,000 mg/m2 IV over 4 hrs, on Days 1, 2, 3, 4, 5. Filgrastim 5 mcg/kg per day SC beginning 24 hrs PRIOR to start of chemotherapy. EPOCH-F: Fludarabine25 mg/m2 per day IV infusion over 30 min., daily on days 1-4. Etoposide 50 mg/m2 per day continuous IV infusion over 24 hrs on days 1-4. Doxorubicin10 mg/m2/d. Grp 2 Alemtuzumab for 4 days starting 8 days before SCT + cyclosporine starting 1 day before SCT and continuing for 6 months.
- Total: Total of all reporting groups
Arm/Group | Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | Cyclosporine (AC) Arm | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 41 | 79
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.92 (14.68) | 47.89 (13.4) | 47.90 (14.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 28 | 30 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 42 | 43 | 85
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 38 | 39 | 77
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44 | 45 | 89
Histology [Count of Participants; unit: Participants] — Acute Myeloid Leukemia (AML)/Myelodysplastic Syndrome (MDS); Cutaneous T Cell Lymphoma (CTCL)/Peripheral T Cell Lymphoma (PTCL)
  Participants
    Non Hodgkin's Lymphoma (NHL) | 11 | 14 | 25
    Hodgkin's Lymphoma (HL) | 5 | 5 | 10
    Chroni Lymphocytic Leukemia (CLL) | 9 | 9 | 18
    AML/MDS | 6 | 5 | 11
    Chronic Myeloid Leukemia (CML) | 4 | 1 | 5
    CTCL/PTCL | 3 | 2 | 5
    Acute Lymphoblastic Leukemia (ALL) | 2 | 2 | 4
    Multiple Myeloma (MM) | 1 | 1 | 2
    Other | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade II-IV Acute Graft Versus Host Disease (GVHD)
Description: Acute GVHD is assessed by the 1994 Consensus Conference on Acute GVHD Grading criteria. See Przepiorka D, Weisdorf D, Martin P, et al. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995; 15:825-8., for grading criteria.
Time Frame: 6 months
Population: 2 of 44 patients who completed the AC arm were transplanted after our cutoff for data analysis and are not included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm: Rituximab:375 mg/m2 IV, day 1 for patients with CD20-positive disease. Allogenic stem cell transplant (ASCT):Conditioning Chemotherapy:Fludarabine:30 mg/m2 per day IV infusion over 30 minutes, daily On days -6, -5, -4, and -3. Cyclophosphamide:1200 mg/m2 per day IV infusion over 2 hours on Days 6, -5, -4, -3.Mesna: 1200 mg/m2 per day IV infusion, Daily on days 6, -5,-4, and -3.Tacrolimus: 0.02 mg/kg, start day 3. Continue IV or PO. Taper will begin at day +63 if no acute GVHD then at day +119 and discontinue at day +180 as tolerated. Methotrexate: 5mg/m2 IV over 15 minutes on days 1, 3, 6, and 11. Sirolimus: 12 mg PO on days -3 to 63, followed by a taper if GVHD does not develop. Sirolimus: 12 mg PO on days -3 to 63, followed by a taper if GVHD does not develop.FLAG: Fludarabine:25 mg/m2 per day IV over 30 minutes, Daily on days 1-5. Cytarabine: 2,000 mg/m2 IV over 4 hours, on Days 1, 2, 3, 4, 5. Filgrastim: 5 mcg/kg per day SC beginning 24 hours PRIOR to initiation of chemotherapy
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
Number analyzed (Participants) | 39 | 42
percentage of participants | 42 [26 to 57] | 38 [23 to 53]

2. Primary Outcome: Percentage of Participants With Chronic Graft Versus Host Disease (cGVHD)
Description: Chronic GVHD is assessed by the 2005 Chronic GVHD Consensus Project. First the individual organ scoring is done, and then based on that the Global score is determined (mild-moderate-severe). See Citation: Filipovich AH, Weisdorf D, Pavletic S, et al. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005; 11:945-56., for grading criteria.
Time Frame: 2 years post transplant
Population: 2 of 44 patients who completed the AC arm were transplanted after our cutoff for data analysis and are not included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
Number analyzed (Participants) | 39 | 42
percentage of participants
  Moderate or Severe cGVHD | 50 [32 to 65] | 12 [4 to 25]
  Severe cGVHD | 28 [14 to 43] | 5 [1 to 15]

3. Primary Outcome: Recovery of Naïve Cluster of Differentiation 4 (CD4) T Cells
Description: The percentage of C-C motif chemokine receptor 7 (CCR7)+CD45RA+ naïve T cells within the CD4 T cell populations was determined by flow cytometry.
Time Frame: Recipient recovery at 6, 12 and 24 months post transplant
Population: A few measurements were missed, one patient was not evaluable for technical reasons and removed from the analysis, but most of the decline was due to patients that had gone off study.
Measure: Median (Full Range); unit: % of naive (CCR7+CD45RA+) CD4 Cells
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
Number analyzed (Participants) | 28 | 28
% of naive (CCR7+CD45RA+) CD4 Cells
  6 mo (TMS=28; AC= 28) | 24 [2 to 65] | 1 [0 to 22]
  12 mo (TMS=25; AC= 21) | 22 [5 to 48] | 7 [0 to 42]
  24 mo (TMS=18; AC= 13) | 20 [4 to 60] | 25 [1 to 60]

4. Primary Outcome: Recovery of Naïve Cluster of Differentiation 8 (CD8) T Cells
Description: The percentage of CCR7+CD45RA+ naïve T cells within the CD4 and CD8 T cell populations was determined by flow cytometry.
Time Frame: Recipient recovery at 6, 12 and 24 months post transplant
Population: as for outcome 3
Measure: Median (Full Range); unit: % of naive (CCR7+CD45RA+) CD8 Cells
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
Number analyzed (Participants) | 28 | 28
% of naive (CCR7+CD45RA+) CD8 Cells
  6 mo (TMS=28; AC= 28) | 20 [0 to 75] | 3 [0 to 78]
  12 mo (TMS=25; AC= 21) | 17 [7 to 79] | 6 [0 to 79]
  24 mo (TMS=18; AC= 13) | 16 [1 to 60] | 6 [0 to 65]

5. Primary Outcome: Changes in Cluster of Differentiation 4 (CD4) T Cell Receptor Vbeta Repertoire
Description: Ribonucleic acid (RNA) was extracted from sorted CD4 and cluster of differentiation 8 (CD8) T cells and analyzed for Vbeta repertoire by nested polymerase chain reaction (PCR) analysis using Vbeta family specific primers and a labeled constant region primer (spectratyping). The receptor repertoire diversity was calculated from spectratyping data by creating a normal standard for repertoire diversity from healthy normal controls and assessing the divergence of individual patient's T cell receptor repertoire from these standard normal donor values. In this Vbeta repertoire divergence index, lower numbers are consistent with a more normal highly diverse repertoire, and high numbers represent a highly skewed, oligoclonal repertoire. The assay is described in Memon SA et al, J Immunol Methods, 2012, 375: 84-92. The repertoire diversity of the CD4 and CD8 T cells of the donor infusion is shown for comparison.
Time Frame: Donor at time of collection and recipient at 1, 3, 6 and 12 months post transplant
Population: The original intention was to perform these assays on the first 10 pts within each arm. One pt died within the first mo., others died within the 1st yr. Not all donors gave consent for research analyses to be done on their cells, hence cells from those donors were not available.
Measure: Median (Full Range); unit: Divergence index
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
Number analyzed (Participants) | 8 | 9
Divergence index
  1 month | 48 [26 to 69] | 90 [63 to 111]
  3 months | 31 [23 to 60] | 66 [47 to 93]
  6 mo (TMS=7; AC= 9) | 35 [21 to 57] | 75 [32 to 93]
  12 mo (TMS=7; AC=9) | 30 [23 to 81] | 67 [25 to 92]
  Donor CD4 cells (TMS=8; AC=8) | 23 [17 to 29] | 22 [18 to 35]

6. Primary Outcome: Changes in CD8 T Cell Receptor Vbeta Repertoire
Description: as for outcome 5
Time Frame: Donor at time of collection and recipient at 1, 3, 6 and 12 months post transplant
Population: as for outcome 5
Measure: Median (Full Range); unit: Divergence index
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
Number analyzed (Participants) | 8 | 9
Divergence index
  1 month | 62 [42 to 91] | 78 [53 to 111]
  3 months | 54 [35 to 64] | 81 [52 to 88]
  6 mo (TMS=7; AC= 9) | 62 [53 to 81] | 84 [71 to 118]
  12 mo (TMS=7; AC= 9) | 55 [39 to 108] | 89 [58 to 110]
  Donor CD8 cells (TMS=8; AC= 8) | 47 [27 to 53] | 43 [31 to 62]

7. Secondary Outcome: Percentage of Participants With Grade III-IV Acute Graft Versus Host Disease (GVHD)
Description: as for outcome 1
Time Frame: 6 months
Population: 2 of 44 patients who completed the AC arm were transplanted after our cutoff for data analysis and are not included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
Number analyzed (Participants) | 39 | 42
percentage of participants | 13 [5 to 26] | 21 [11 to 35]

8. Secondary Outcome: Toxicities
Description: Here are the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 103 months and 22 days
Measure: Number; unit: participants
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
Number analyzed (Participants) | 44 | 45
participants | 43 | 42

9. Secondary Outcome: Days to Engraftment of Neutrophils
Description: Days to engraftment is defined as neutrophil recovery: designated by the first of 3 consecutive days with an absolute neutrophil count (ANC) above 500/mm(3).
Time Frame: 2 years
Population: One myeloma patient had graft failure in the AC Arm. 2 of 44 patients who completed the AC arm were transplanted after our cutoff for data analysis and are not included.
Measure: Median (Full Range); unit: Days to neutrophil engraftment
Groups:
- B - Cyclosporine (AC Arm): Rituximab375 mg/m2 IV, day 1 for pts with CD20-positive disease. Cyclosporine IV over 2 hrs or orally every 12 hrs on days -1-100, followed by a taper if GVHD does not develop. Allogenic stem cell transplant. Conditioning Chemotherapy Fludarabine:30 mg/m2 per day IV infusion over 30 min., daily on days -6, -5, -4, and -3. Cyclophosphamide1200 mg/m2 per day IV infusion over 2 hrs on Days 6, -5, -4, -3. Mesna1200 mg/m2 per day IV infusion, Daily on days 6, -5,-4, and -3. FLAG: Fludarabine25 mg/m2 per day IV over 30 min., Daily on days 1-5. Cytarabine 2,000 mg/m2 IV over 4 hrs, on Days 1, 2, 3, 4, 5. Filgrastim 5 mcg/kg per day SC beginning 24 hrs PRIOR to start of chemotherapy. EPOCH-F: Fludarabine25 mg/m2 per day IV infusion over 30 min., daily on days 1-4. Etoposide 50 mg/m2 per day continuous IV infusion over 24 hrs on days 1-4. Doxorubicin10 mg/m2/d. Grp 2 Alemtuzumab for 4 days starting 8 days before SCT + cyclosporine starting 1 day before SCT and continuing for 6 months.
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC Arm)
Number analyzed (Participants) | 39 | 42
Days to neutrophil engraftment | 11 [3 to 19] | 9 [7 to 36]

10. Secondary Outcome: Days to Engraftment of Platelets
Description: Platelet recovery: designated by the first of 7 days where the platelet count remains above 20,000/mm(3) without transfusion support
Time Frame: 2 years
Population: 2 of 44 patients who completed the AC arm were transplanted after our cutoff for data analysis and are not included.
Measure: Median (Full Range); unit: Days
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC Arm)
Number analyzed (Participants) | 39 | 42
Days | 19 [1 to 99] | 14 [1 to 431]

11. Secondary Outcome: Days to Engraftment of Lymphocytes
Description: Lymphocyte recovery: designated by the first of 3 consecutive days with absolute lymphocyte count (ALC) above 500/mm(3).
Time Frame: 2 years
Population: 2 of 44 patients who completed the AC arm were transplanted after our cutoff for data analysis and are not included.
Measure: Median (Full Range); unit: Days
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC Arm)
Number analyzed (Participants) | 39 | 42
Days | 16 [1 to 194] | 76 [16 to 264]

12. Secondary Outcome: Overall Survival
Description: Time between the first day of transplant to the day of death.
Time Frame: Patients were followed for an average of up to 5 years.
Population: 2 of 44 patients who completed the AC arm were transplanted after our cutoff for data analysis and are not included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
Number analyzed (Participants) | 39 | 42
Months | 41.7 [26.7 to NA] — The upper limit is undefined because there are too few deaths for it to be determined. | 18.8 [10.4 to NA] — The upper limit is undefined because there are too few deaths for it to be determined.

13. Secondary Outcome: Early Treatment Related Mortality
Description: Any death occurring within 28 days after transplantation in a patient in continuous remission.
Time Frame: Less than or equal to 28 days after transplantation
Population: 2 of 44 patients who completed the AC arm were transplanted after our cutoff for data analysis and are not included.
Measure: Number; unit: participants
Groups:
- B - Cyclosporine (C) Arm: Rituximab375 mg/m2 IV, day 1 for pts with CD20-positive disease. Cyclosporine IV over 2 hrs or orally every 12 hrs on days -1-100, followed by a taper if GVHD does not develop. Allogenic stem cell transplant. Conditioning Chemotherapy Fludarabine:30 mg/m2 per day IV infusion over 30 min., daily on days -6, -5, -4, and -3. Cyclophosphamide1200 mg/m2 per day IV infusion over 2 hrs on Days 6, -5, -4, -3. Mesna1200 mg/m2 per day IV infusion, Daily on days 6, -5,-4, and -3. FLAG: Fludarabine25 mg/m2 per day IV over 30 min., Daily on days 1-5. Cytarabine 2,000 mg/m2 IV over 4 hrs, on Days 1, 2, 3, 4, 5. Filgrastim 5 mcg/kg per day SC beginning 24 hrs PRIOR to start of chemotherapy. EPOCH-F: Fludarabine25 mg/m2 per day IV infusion over 30 min., daily on days 1-4. Etoposide 50 mg/m2 per day continuous IV infusion over 24 hrs on days 1-4. Doxorubicin10 mg/m2/d. Grp 2 Alemtuzumab for 4 days starting 8 days before SCT + cyclosporine starting 1 day before SCT and continuing for 6 months.
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (C) Arm
Number analyzed (Participants) | 39 | 42
participants | 1 | 0

14. Secondary Outcome: Percentage of Participants With Late Treatment Related Mortality
Description: Any death occurring 28 days or more after transplantation in a patient in continuous remission.
Time Frame: Greater than 28 days after transplantation
Population: 2 of 44 patients who completed the AC arm were transplanted after our cutoff for data analysis and are not included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
Number analyzed (Participants) | 39 | 42
percentage of participants | 28 [14 to 43] | 29 [16 to 44]

15. Secondary Outcome: Decline in Homeostatic Cytokine Interleukin 7 (IL-7) Post-Transplant
Description: During depletion of lymphocytes during transplant conditioning, levels of homeostatic cytokines increase in the blood. These then decline with the expansion of new donor-derived cells. The rapidity of decline may predict acute graft versus host disease (AGVHD). Decline in cytokine IL-7 will be assessed by the enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 0, 1 week and 2 weeks
Population: Following the focus on chronic graft-versus host disease (GVHD) as a primary outcome measure in 2011, this measure was not assessed.
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (C) Arm
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Immune Reconstitution of Normal Killer (NK) Cells
Description: Cluster of differentiation 3 (CD3) - cluster of differentiation 56 (CD56) + Natural Killer (NK) cells within the lymphocyte population were determined by flow cytometry. The absolute numbers of cells/µl were calculated from the absolute lymphocyte count.
Time Frame: 2 weeks, and 1, 3, 6, 12, and 24 months post transplant
Population: 2 of 44 patients who completed the AC arm were transplanted after our cutoff for data analysis and are not included. A total of 5 completed participants did not contribute data due to missing samples, and participants who died and were not able to supply samples for the time points indicated.
Measure: Median (Full Range); unit: Cells/µl
Groups:
- A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm: TMS Arm Rituximab: 375 mg/m2 IV, day 1 for patients with cluster of differentiation 20 (CD20)-positive disease Allogenic stem cell transplant (ASCT):Allogenic stem cell transplant Conditioning Chemotherapy:Fludarabine:30 mg/m2 per day IV infusion over 30 minutes, daily. On days -6, -5, -4, and -3 Cyclophosphamide:1200 mg/m2 per day IV infusion over 2 hours on Days 6, -5, -4, -3 Mesna:1200 mg/m2 per day IV infusion, Daily on days 6, -5,-4, and -3 TMS: Tacrolimus: 0.02 mg/kg, start day 3. Continue IV or PO. Taper will begin at day +63 if no acute GVHD then at day +119 and discontinue at day +180 as tolerated Methotrexate: 5 mg/m2 IV over 15 minutes on days 1, 3, 6, and 11 Sirolimus: 12 mg PO on days -3 to 63, followed by a taper if GVHD does not develop.
  FLAG: Fludarabine:25 mg/m2 per day IV over 30 minutes, Daily on days 1-5 Cytarabine: 2,000 mg/m2 IV over 4 hours, on Days 1, 2, 3, 4, 5 Filgrastim: 5 mcg/kg per day SC beginning 24 hours PRIOR to initiation of chemotherapy
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
Number analyzed (Participants) | 38 | 39
Cells/µl
  2 weeks: number analyzed (Participants) | 36 | 39
  2 weeks | 123 [5 to 538] | 15 [0 to 331]
  1 month: number analyzed (Participants) | 38 | 37
  1 month | 270 [41 to 940] | 31 [0 to 936]
  3 months: number analyzed (Participants) | 34 | 34
  3 months | 134 [22 to 575] | 124 [1 to 794]
  6 months: number analyzed (Participants) | 30 | 28
  6 months | 136 [25 to 442] | 202 [1 to 831]
  12 months: number analyzed (Participants) | 25 | 24
  12 months | 134 [12 to 366] | 150 [16 to 1043]
  24 months: number analyzed (Participants) | 22 | 17
  24 months | 133 [27 to 798] | 307 [133 to 1336]

17. Secondary Outcome: Immune Reconstitution of Cluster of Differentiation 4 (CD4) T Cell Populations
Description: Cluster of Differentiation 3 (CD3)+CD4+ and CD3+Cluster of Differentiation 8 (CD8)+ T cells within the lymphocyte population were determined by flow cytometry. The absolute numbers of cells/µl were calculated from the absolute lymphocyte count.
Time Frame: 2 weeks, and 1, 3, 6, 12 and 24 months post transplant
Population: as for outcome 16
Measure: Median (Full Range); unit: Cells/µl
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
Number analyzed (Participants) | 38 | 39
Cells/µl
  2 weeks: number analyzed (Participants) | 36 | 39
  2 weeks | 171 [14 to 536] | 0 [0 to 131]
  1 month: number analyzed (Participants) | 38 | 37
  1 month | 285 [15 to 2816] | 21 [0 to 276]
  3 months: number analyzed (Participants) | 34 | 34
  3 months | 297 [3 to 1178] | 61 [9 to 1109]
  6 months: number analyzed (Participants) | 30 | 28
  6 months | 387 [79 to 1126] | 121 [26 to 2201]
  12 months: number analyzed (Participants) | 25 | 24
  12 months | 447 [55 to 1821] | 132 [7 to 619]
  24 months: number analyzed (Participants) | 22 | 17
  24 months | 451 [143 to 893] | 373 [64 to 1765]

18. Secondary Outcome: Immune Reconstitution of Cluster of Differentiation 8 (CD8) T Cell Populations
Description: Cluster of differentiation 3 (CD3)+cluster of differentiation 4 (CD4)+ and CD3+CD8+ T cells within the lymphocyte population were determined by flow cytometry. The absolute numbers of cells/µl were calculated from the absolute lymphocyte count.
Time Frame: 2 weeks, 1, 3, 6, 12 and 24 months post transplant
Population: as for outcome 16
Measure: Median (Full Range); unit: Cells/µl
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
Number analyzed (Participants) | 38 | 39
Cells/µl
  2 weeks: number analyzed (Participants) | 36 | 39
  2 weeks | 72 [9 to 560] | 1 [0 to 240]
  1 month: number analyzed (Participants) | 38 | 37
  1 month | 204 [10 to 2147] | 6 [0 to 430]
  3 months: number analyzed (Participants) | 34 | 34
  3 months | 334 [3 to 1054] | 54 [1 to 846]
  6 months: number analyzed (Participants) | 30 | 28
  6 months | 429 [79 to 1487] | 158 [0 to 1302]
  12 months: number analyzed (Participants) | 25 | 24
  12 months | 485 [64 to 1844] | 243 [1 to 2861]
  24 months: number analyzed (Participants) | 22 | 17
  24 months | 434 [121 to 1928] | 502 [92 to 4239]

ADVERSE EVENTS:
Time Frame: 103 months and 22 days
Description: One participant was enrolled and given induction chemotherapy but was never randomized to Arm TMS or AC. Subject had one AE (infection with normal ANC or Grade 1 or 2 neutrophils: Pharynx). Subject was taken off study for disease progression and died.
Groups:
- A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm: TMS Arm
  Rituximab: Rituximab: 375 mg/m2 IV, day 1 for patients with CD20-positive disease
  Allogenic stem cell transplant (ASCT): Allogenic stem cell transplant
  Conditioning Chemotherapy: Fludarabine:30 mg/m2 per day IV infusion over 30 minutes, daily On days -6, -5, -4, and -3 Cyclophosphamide:1200 mg/m2 per day IV infusion over 2 hours on Days 6, -5, -4, -3 Mesna: 1200 mg/m2 per day IV infusion, Daily on days 6, -5,-4, and -3
  TMS: Tacrolimus: 0.02 mg/kg , start day 3. Continue IV or PO. Taper will begin at day +63 if no acute GVHD then at day +119 and discontinue at day +180 as tolerated Methotrexate: 5 mg/m2 IV over 15 minutes on days 1, 3, 6, and 11. Sirolimus: 12 mg PO on days -3 to 63, followed by a taper if GVHD does not develop.
  FLAG: Fludarabine:25 mg/m2 per day IV over 30 minutes, Daily on days 1-5 Cytarabine: 2,000 mg/m2 IV over 4 hours,on Days 1, 2, 3, 4, 5 Filgrastim: 5 mcg/kg per day SC beginning 24 hours PRIOR to initiation of chemotherapy
- B - Cyclosporine (AC) Arm: AC Arm
  Rituximab: Rituximab: 375 mg/m2 IV, day 1 for patients with CD20-positive disease
  Cyclosporine: Cyclosporine: IV over 2 hours or orally every 12 hours on days -1 to 100, followed by a taper if GVHD does not develop.
  Allogenic stem cell transplant (ASCT): Allogenic stem cell transplant
  Conditioning Chemotherapy: Fludarabine:30 mg/m2 per day IV infusion over 30 minutes, daily On days -6, -5, -4, and -3 Cyclophosphamide:1200 mg/m2 per day IV infusion over 2 hours on Days 6, -5, -4, -3 Mesna: 1200 mg/m2 per day IV infusion, Daily on days 6, -5,-4, and -3
  FLAG: Fludarabine:25 mg/m2 per day IV over 30 minutes, Daily on days 1-5 Cytarabine: 2,000 mg/m2 IV over 4 hours,on Days 1, 2, 3, 4, 5 Filgrastim: 5 mcg/kg per day SC beginning 24 hours PRIOR to initiation of chemotherapy EPOCH-F: Fludarabine:25 mg/m2 per day IV infusion over 30 minutes, daily on days 1-4 Etoposide :50 mg/m2 per day continuous IV infusion over 24 hours on days 1-4 Doxorubicin:10 mg/m2/d
Arm/Group | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm | B - Cyclosporine (AC) Arm
All-Cause Mortality (participants affected / at risk) | 8/44 | 19/45
Serious Adverse Events (participants affected / at risk) | 36/44 | 41/45
Other Adverse Events (participants affected / at risk) | 43/44 | 42/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm (N=44) | B - Cyclosporine (AC) Arm (N=45)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 4 (5) | 1 (2)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 4 (6) | 1 (2)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2) | 0 (0)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ataxia (incoordination) (Nervous system disorders) | 0 (0) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 1 (1)
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary arrest, cause unknown (non-fatal) (Cardiac disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Gastrointestinal disorders) | 5 (8) | 7 (12)
Confusion (Nervous system disorders) | 1 (1) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 3 (5) | 2 (3)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 0 (0) | 1 (1)
Death not associated with CTCAE term::Death NOS (General disorders) | 4 (4) | 7 (7)
Death not associated with CTCAE term::Disease progression NOS (General disorders) | 3 (3) | 10 (10)
Death not associated with CTCAE term::Multi-organ failure (General disorders) | 1 (1) | 2 (2)
Dermatology/Skin - Other (Deep sclerosis per MRI, GVHD possible) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 8 (9) | 8 (10)
Dry eye syndrome (Eye disorders) | 3 (3) | 0 (0)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Edema: limb (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Edema: viscera (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 3 (3)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Infections and infestations) | 6 (7) | 6 (9) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (2) | 1 (1)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 3 (10) | 2 (4)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemorrhage, CNS (Nervous system disorders) | 0 (0) | 2 (2)
Hemorrhage, GI::Abdomen NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GI::Duodenum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GI::Lower GI NOS (Gastrointestinal disorders) | 0 (0) | 3 (3)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GI::Upper GI NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, pulmonary/upper respiratory::Lung (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 5 (5)
Hypotension (Cardiac disorders) | 3 (4) | 5 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 8 (13)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1) | 1 (1)
Infection:: Abdomen NOS (Infections and infestations) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::
Infection ::Bladder (urinary) (Infections and infestations) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection ::Blood (Infections and infestations) | 3 (3) | 8 (10) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection::Catheter-related (Infections and infestations) | 1 (1) | 4 (5) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection ::Lip/perioral (Infections and infestations) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection ::Lung (pneumonia) (Infections and infestations) | 4 (6) | 3 (3) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection::Meninges (meningitis) (Infections and infestations) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection ::Muscle (infection myositis) (Infections and infestations) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection::Nose (Infections and infestations) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection::Rectum (Infections and infestations) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection::Sinus (Infections and infestations) | 2 (2) | 2 (2) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection ::Trachea (Infections and infestations) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection::Upper airway NOS (Infections and infestations) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection ::Urinary tract NOS (Infections and infestations) | 2 (2) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection - Other (Infections and infestations) | 1 (3) | 2 (3) — (S. Aureus positive blood; gram-neg-rod; line infection)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bladder (urinary) (Infections and infestations) | 1 (1) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 9 (15) | 21 (40)
Infection with normal ANC or Grade 1 or 2 neutrophils::Brain (encephalitis, infectious) (Infections and infestations) | 3 (3) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bronchus (Infections and infestations) | 2 (3) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Catheter-related (Infections and infestations) | 4 (4) | 12 (14)
Infection with normal ANC or Grade 1 or 2 neutrophils::Colon (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Esophagus (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Heart (endocarditis) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Liver (Infections and infestations) | 1 (1) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 10 (18) | 13 (30)
Infection with normal ANC or Grade 1 or 2 neutrophils::Meninges (meningitis) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Paranasal (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Pharynx (Infections and infestations) | 2 (2) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Sinus (Infections and infestations) | 4 (4) | 6 (8)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 2 (3) | 4 (5)
Infection with normal ANC or Grade 1 or 2 neutrophils::Stomach (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 1 (1) | 3 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils::Wound (Infections and infestations) | 1 (1) | 1 (1)
Infection with unknown ANC::Blood (Infections and infestations) | 2 (2) | 2 (2)
Infection with unknown ANC::Catheter-related (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC::Colon (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 2 (2) | 1 (1)
Iron overload (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 2 (3) | 4 (4)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
Leukoencephalopathy (radiographic findings) (Nervous system disorders) | 0 (0) | 1 (1)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 3 (3) | 0 (0)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — (sclerodermic & fascial changes; leg cramping/edema possible GVHD, prednisone started)
Myositis (inflammation/damage of muscle) (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3 (4) | 1 (3)
Ocular/Visual - Other (Eye disorders) | 0 (0) | 1 (1) — (idiopathic progressive retinal vasculitis; poss inflammatory process; uk etiology; total blindness)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain::Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain::Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pancreatic endocrine: glucose intolerance (Endocrine disorders) | 2 (2) | 1 (1)
Perforation, GI::Small bowel NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pericardial effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (2) | 2 (11)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (5)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, respiratory failure) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory - Other (pleural thickening) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (5) | 7 (10)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 10 (12) | 6 (10)
Renal/Genitourinary - Other (AKI, required CVVH) (Renal and urinary disorders) | 0 (0) | 1 (1)
Right ventricular dysfunction (cor pulmonale) (Cardiac disorders) | 0 (0) | 1 (1)
Secondary Malignancy - possibly related to cancer treatment (AML); (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (5) — possibly related to cancer treatment (PTLD(liver biopsy + 10/3/08, stomach bx 10/6/08), EBV associated; to cancer treatment (EBV associated PTLD, neck LN bx (+)10/12/11;to cancer treatment (EBV assoc. PTLD;tonsil bx 10/12/11;obstructing nasopharynx).
Secondary Malignancy - possibly related to cancer treatment (metastat. test cancer in lung) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Stricture/stenosis (including anastomotic), GI::Esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia::Atrial fibrillation (Cardiac disorders) | 3 (5) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Supraventricular and nodal arrhythmia::Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 2 (2) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 4 (5) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1) — (e.g., thrombotic thrombocytopenic purpura [TTP] or hemolytic uremic syndrome [HUS])
Tumor lysis syndrome (General disorders) | 0 (0) | 1 (1)
Ulcer, GI::Duodenum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia::Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Weight gain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - Tacrolimus, Methotrexate, Sirolimus (TMS) Arm (N=44) | B - Cyclosporine (AC) Arm (N=45)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 28 (75) | 17 (45)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 26 (73) | 23 (50)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 9 (15) | 12 (23)
Alkaline phosphatase (Metabolism and nutrition disorders) | 7 (20) | 6 (9)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0)
Amylase (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Anorexia (Gastrointestinal disorders) | 2 (2) | 2 (4)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 12 (22) | 16 (38)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 1 (4) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Cardiac General - Other (cardimyopathy) (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac General - Other (heart failure, fluid overload) (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Colitis, infectious (e.g., Clostridium difficile) (Gastrointestinal disorders) | 1 (1) | 2 (2)
Confusion (Nervous system disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 9 (11) | 10 (16)
Cystitis (Renal and urinary disorders) | 1 (1) | 1 (1)
Dermatology/Skin - Other (GVHD; cGVHD) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatology/Skin - Other (MRSA abscess) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 20 (25) | 22 (32)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 8 (8) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 3 (4) | 1 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Edema: head and neck (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
FEV(1) (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2) | 5 (5)
Febrile neutropenia (Infections and infestations) | 4 (4) | 9 (9) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (Infections and infestations) | 3 (3) | 9 (12)
Fibrinogen (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fistula, GI::Anus (Gastrointestinal disorders) | 1 (1) | 0 (0)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal - Other (GVHD) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal - Other (Gastrointestinal disorders) | 0 (0) | 1 (1) — (duodenal bx 1/24/11; very rare apoptotic cells CMV stains (-); steroids started for GVHD)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 26 (108) | 26 (150)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Hemorrhage, GI::Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI::Anus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI::Lower GI NOS (Gastrointestinal disorders) | 1 (3) | 0 (0)
Hemorrhage, GU::Bladder (Renal and urinary disorders) | 3 (3) | 0 (0)
Hemorrhage, GU::Urinary NOS (Renal and urinary disorders) | 0 (0) | 1 (1)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Hypertension (Cardiac disorders) | 3 (3) | 7 (7)
Hypotension (Cardiac disorders) | 2 (2) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (8)
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (2) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Abdomen NOS
Infection ::Bladder (urinary) (Infections and infestations) | 6 (6) | 3 (3) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection::Blood (Infections and infestations) | 9 (12) | 11 (14) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection::Brain (encephalitis, infectious) (Infections and infestations) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection ::Brain + Spinal cord (encephalomyelitis) (Infections and infestations) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection::Bronchus (Infections and infestations) | 2 (2) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection ::Catheter-related (Infections and infestations) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection ::Colon (Infections and infestations) | 2 (2) | 3 (3) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection ::Eye NOS (Infections and infestations) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection ::Lip/perioral (Infections and infestations) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection ::Lung (pneumonia) (Infections and infestations) | 6 (8) | 6 (6) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection::Oral cavity-gums (gingivitis) (Infections and infestations) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection Sinus (Infections and infestations) | 2 (2) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::
Infection::Skin (cellulites) (Infections and infestations) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection::Soft tissue NOS (Infections and infestations) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L
Infection ::Upper aerodigestive NOS (Infections and infestations) | 1 (1) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection:: Upper airway NOS (Infections and infestations) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection::Urinary tract NOS (Infections and infestations) | 2 (2) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection ::Wound (Infections and infestations) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection - Other (CMV reactivation) (Infections and infestations) | 0 (0) | 1 (1)
Infection - Other (Rhinovirus, Coronavirus HKU1) (Infections and infestations) | 0 (0) | 1 (1)
Infection - Other (Varicella zoster; noravirus) (Infections and infestations) | 2 (2) | 0 (0)
Infection - Other (acinetobacter) (Infections and infestations) | 0 (0) | 1 (1)
Infection - Other (dissiminated HSV) (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bladder (urinary) (Infections and infestations) | 3 (3) | 4 (5)
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 20 (44) | 25 (62)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bronchus (Infections and infestations) | 1 (1) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils::Catheter-related (Infections and infestations) | 0 (0) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Colon (Infections and infestations) | 2 (2) | 2 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils::Conjunctiva (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Eye NOS (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 7 (8) | 12 (18)
Infection with normal ANC or Grade 1 or 2 neutrophils::Nose (Infections and infestations) | 2 (3) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Paranasal (Infections and infestations) | 0 (0) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Penis (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Pharynx (Infections and infestations) | 2 (2) | 3 (5)
Infection with normal ANC or Grade 1 or 2 neutrophils::Sinus (Infections and infestations) | 4 (6) | 9 (10)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 2 (2) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils::Stomach (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Trachea (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper aerodigestive NOS (Infections and infestations) | 1 (1) | 2 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 9 (14) | 9 (10)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 4 (4) | 5 (6)
Infection with normal ANC or Grade 1 or 2 neutrophils::Vagina (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Wound (Infections and infestations) | 0 (0) | 3 (4)
Infection with unknown ANC::Blood (Infections and infestations) | 4 (4) | 2 (3)
Infection with unknown ANC::Bronchus (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC::Catheter-related (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 1 (1) | 1 (1)
Infection with unknown ANC::Sinus (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC::Skin (cellulites) (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC::Upper aerodigestive NOS (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC::Upper airway NOS (Infections and infestations) | 6 (7) | 2 (2)
Infection with unknown ANC::Urinary tract NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC::Wound (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0)
Iron overload (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Joint-function (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 27 (118) | 26 (189)
Leukoencephalopathy (radiographic findings) (Nervous system disorders) | 0 (0) | 1 (1)
Lipase (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 27 (143) | 27 (181)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 13 (22) | 16 (26)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 (4) | 9 (15)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic/Laboratory - Other (pancytopenia; steroid induced hyperglycemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Mood alteration::Anxiety (Nervous system disorders) | 2 (2) | 2 (2)
Mood alteration::Depression (Nervous system disorders) | 1 (1) | 3 (3)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 10 (10) | 0 (0)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 8 (8) | 2 (2)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-lower (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 16 (17) | 6 (7)
Neurology - Other (delirium) (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 2 (2) | 2 (2)
Neuropathy: sensory (Nervous system disorders) | 4 (4) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 26 (109) | 27 (123)
Obstruction, GU::Bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1 (1) | 0 (0)
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 0 (0) | 1 (1)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 5 (5) | 8 (15)
Pain::Anus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pain::Back (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 2 (2) | 2 (2)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain::Throat/pharynx/larynx (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain::Urethra (Renal and urinary disorders) | 1 (1) | 0 (0)
Pancreatic endocrine: glucose intolerance (Endocrine disorders) | 3 (3) | 1 (1)
Perforation, GI::Small bowel NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pericardial effusion (non-malignant) (Cardiac disorders) | 2 (2) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 20 (69) | 22 (53)
Platelets (Blood and lymphatic system disorders) | 25 (81) | 23 (106)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (3) | 10 (15)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 10 (16) | 17 (36)
Prolonged QTc interval (Cardiac disorders) | 1 (1) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory - Other (infiltrates) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) — Infiltrates; fungal pneumonia
Pulmonary/Upper Respiratory - Other (infiltrates; fungal pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 19 (30) | 26 (39)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (5) | 4 (4)
Renal/Genitourinary - Other (acute renal injury) (Renal and urinary disorders) | 3 (4) | 0 (0) — dysuria; hematuria; stent replacement; fluid overload refractory to normal doses of Lasix
Renal/Genitourinary - Other (dysuria) (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (dysuria; hematuria; stent replacement) (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (failure; hematuria; insufficiency; dysuria) (Renal and urinary disorders) | 0 (0) | 6 (7)
Renal/Genitourinary - Other (fluid overload refractory to normal doses of Lasix) (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (hematuria) (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (insufficiency) (Renal and urinary disorders) | 4 (4) | 0 (0)
Right ventricular dysfunction (cor pulmonale) (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Rigors/chills (General disorders) | 0 (0) | 1 (1)
Secondary Malignancy - possibly related to cancer treatment (mucoepidermoid carcinoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Secondary Malignancy - possibly related to cancer treatment (squamous cell carcinoma lip) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Skin breakdown/decubitus ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 6 (9) | 9 (11)
Supraventricular and nodal arrhythmia::Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 1 (1)
Syndromes - Other (septic shock) (General disorders) | 0 (0) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1) | 2 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 6 (6) | 2 (2)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 4 (4) — (e.g., thrombotic thrombocytopenic purpura [TTP] or hemolytic uremic syndrome [HUS])
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 0 (0) | 1 (1)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 4 (5) | 7 (16)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Vaginal mucositis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Weight loss (General disorders) | 1 (1) | 0 (0)
Wound complication, non-infectious (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT00520130/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT00520130/ICF_001.pdf